CLINICAL TRIAL: NCT01412957
Title: A Phase 3, Multicenter, Randomized, Open-label Trial to Evaluate the Survival Benefit of Panitumumab and Best Supportive Care, Compared to Best Supportive Care Alone, in Subjects With Chemorefractory Wild-type KRAS Metastatic Colorectal Cancer
Brief Title: Comparison of Survival Benefit of Panitumumab With Supportive Care to Best Supportive Care Alone in Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20100007; 2010-022951-49 (EudraCT Number)
Record Dates: First submitted 2011-03-31; First posted 2011-08-09 (Estimated); Results first posted 2016-04-08 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-02

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Best Supportive Care; Panitumumab; Chemorefractory; Wild-type KRAS; Overall Survival; Phase 3
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Panitumumab + BSC (Experimental): Participants received panitumumab administered intravenously 6 mg/kg every 14 days plus BSC until disease progression, withdrawal of consent, death, or intolerance of study drug.
  Interventions: Other: Best Supportive Care (BSC); Drug: Panitumumab
- BSC Alone (Other): Participants received best supportive care until disease progression, withdrawal of consent, or death.
  Interventions: Other: Best Supportive Care (BSC)

INTERVENTIONS:
Other: Best Supportive Care (BSC) — BSC was defined as the best palliative care available as judged appropriate by the investigator and according to institutional guidelines and could include antibiotics, analgesics, radiation therapy for pain control (limited to bone metastases), corticosteroids, transfusions, psychotherapy, growth factors, palliative surgery, or any other symptomatic therapy as clinically indicated.
Drug: Panitumumab — Administered intravenously
  Other Names: Vectibix
  Arms: Panitumumab + BSC

SUMMARY:
The purpose of this study is to evaluate the benefit of panitumumab in addition to best supportive care compared to best supportive care alone in patients with chemorefractory wild-type KRAS (Kirsten rat sarcoma viral oncogene homolog) metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of metastatic colorectal cancer (CRC)
* Wild-type (without mutation in codons 12 and 13) KRAS gene in tumor tissue confirmed by a central laboratory
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* At least 1 measurable or non-measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 guidelines.
* Treatment failure (defined as failure due to either disease progression [clinical or radiological] or toxicity [treatment intolerance]) of a prior regimen containing irinotecan for metastatic disease and a prior regimen containing oxaliplatin for metastatic disease. Oxaliplatin and irinotecan may have been administered sequentially or in combination.

  * Disease relapse within 6 months after completing adjuvant chemotherapy (with either an irinotecan or oxaliplatin containing regimen) will also be considered as treatment failure of a prior regimen for metastatic disease
* Must have previously received a thymidylate synthase inhibitor (eg, fluorouracil, capecitabine, raltitrexed, or fluorouracil-uracil) at any point for treatment of CRC
* Man or woman at least 18 years of age
* Adequate hematologic, renal, hepatic and metabolic function
* Negative pregnancy test within 72 hours before randomization (for women of childbearing potential only)
* Subject or subject's legally acceptable representative has provided informed consent.
* Other protocol-specified criteria may apply

Exclusion Criteria:

* Symptomatic brain metastases requiring treatment
* History of another primary cancer within 5 years of randomization
* Prior anti-epidermal growth factor receptor (EGFR) antibody therapy (eg, panitumumab or cetuximab) or treatment with small molecule EGFR inhibitors (eg, gefitinib, erlotinib, lapatinib)
* Antitumor therapy (eg, chemotherapy, hormonal therapy, immunotherapy, antibody therapy) within 21 days before randomization
* Radiotherapy within 14 days before randomization.
* Exclusion Criteria for corrected QT (QTc) Evaluation Subpart of the Study: Prolongation of QT/QTc interval > 450 milliseconds at screening
* Other protocol-specified criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 377 (Actual)
Dates: Start 2011-11; Primary Completion 2014-06 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (62):
- Brazil (4):
  - Research Site, Curitiba, Paraná
  - Research Site, Natal, Rio Grande do Norte
  - Research Site, Ijuí, Rio Grande do Sul
  - Research Site, Porto Alegre, Rio Grande do Sul
- Canada (4):
  - Research Site, Greenfield Park, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Trois-Rivières, Quebec
- Chile (2):
  - Research Site, Temuco, Cautín
  - Research Site, Viña del Mar, Región de Valparaíso
- China (9):
  - Research Site, Fuzhou, Fujian
  - Research Site, Shijiazhuang, Hebei
  - Research Site, Nanjing, Jiangsu
  - Research Site, Changchun, Jilin
  - Research Site, Shenyang, Liaoning
  - Research Site, Xi'an, Shaanxi
  - Research Site, Beijing
  - Research Site, Chongqing
  - Research Site, Shanghai
- Croatia (5):
  - Research Site, Osijek
  - Research Site, Pula
  - Research Site, Rijeka
  - Research Site, Split
  - Research Site, Zagreb
- Estonia (2):
  - Research Site, Tallinn
  - Research Site, Tartu
- Greece (2):
  - Research Site, Athens
  - Research Site, Chania
- India (8):
  - Research Site, Hyderabad, Andhra Pradesh
  - Research Site, Visakhapatnam, Andhra Pradesh
  - Research Site, Bangalore, Karnataka
  - Research Site, Kochi, Kerala
  - Research Site, Mumbai, Maharashtra
  - Research Site, Nashik, Maharashtra
  - Research Site, Pune, Maharashtra
  - Research Site, Chennai, Tamil Nadu
- Latvia (2):
  - Research Site, Daugavpils
  - Research Site, Riga
- Lithuania (2):
  - Research Site, Kaunas
  - Research Site, Vilnius
- Malaysia (3):
  - Research Site, Kuala Lumpur, Kuala Lumpur
  - Research Site, Kampung Baharu Nilai, Negeri Sembilan
  - Research Site, George Town, Pulau Pinang
- Mexico (3):
  - Research Site, Mexico City, Mexico City
  - Research Site, Cuernavaca, Morelos
  - Research Site, Oaxaca City, Oaxaca
- Philippines (4):
  - Research Site, Davao City, Davao Region
  - Research Site, Cebu City
  - Research Site, Manila
  - Research Site, Pasay
- Romania (7):
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Craiova
  - Research Site, Lasi
  - Research Site, Ploieşti
  - Research Site, Suceava
  - Research Site, Timișoara
- Serbia (3):
  - Research Site, Belgrade
  - Research Site, Kamenitz
  - Research Site, Niš
- South Korea (2):
  - Research Site, Goyang-si, Gyeonggi-do
  - Research Site, Seoul

REFERENCES:
- [Background] Kim TW, Elme A, Kusic Z, Park JO, Udrea AA, Kim SY, Ahn JB, Valencia RV, Krishnan S, Bilic A, Manojlovic N, Dong J, Guan X, Lofton-Day C, Jung AS, Vrdoljak E. A phase 3 trial evaluating panitumumab plus best supportive care vs best supportive care in chemorefractory wild-type KRAS or RAS metastatic colorectal cancer. Br J Cancer. 2016 Nov 8;115(10):1206-1214. doi: 10.1038/bjc.2016.309. Epub 2016 Oct 13. PMID 27736842
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 377 participants were randomized at 66 centers in Europe, Asia, North and South America from 8 November 2011 until 30 July 2013.
  Results are reported as of the primary analysis data cut-off date of 10 June 2014.
Pre-assignment Details: Participants were stratified according to geographic region (Europe vs Asia vs rest of the world) and Eastern Cooperative Oncology Group (ECOG) performance status (0 or 1 vs 2) and randomized (1:1 ratio) to 1 of 2 treatment groups.
Groups:
- Panitumumab + BSC: Participants received panitumumab administered intravenously 6 mg/kg every 14 days plus best supportive care (BSC) until disease progression, withdrawal of consent, death, or intolerance of study drug.
Period: Overall Study
Arm/Group | Panitumumab + BSC | BSC Alone
Started | 189 | 188
Completed | 40 (Participants continuing study at the time of data cut-off) | 31 (Participants continuing study at the time of data cut-off)
Not Completed | 149 | 157
Not completed — Withdrawal by Subject | 6 | 22
Not completed — Lost to Follow-up | 7 | 2
Not completed — Death | 136 | 133

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Panitumumab + BSC | BSC Alone | Total
Number analyzed (Participants) | 189 | 188 | 377
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (10.7) | 58.7 (11.1) | 59.4 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 79 | 161
  Male | 107 | 109 | 216
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 23 | 22 | 45
  Not Hispanic or Latino | 166 | 166 | 332
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 3 | 3
  Asian | 79 | 82 | 161
  White | 107 | 102 | 209
  Other | 3 | 1 | 4
Geographic Region [Number; unit: participants]
  Europe | 86 | 85 | 171
  Asia | 80 | 82 | 162
  Rest of world | 23 | 21 | 44
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — A scale to assess a patient's disease status. 0 = Fully active, able to carry out all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity, ambulatory and able to carry out work of a light nature; 2 = Ambulatory and capable of all self care, unable to carry out any work activities. Up and about > 50% of waking hours; 3 = Capable of only limited self-care, confined to bed or chair > 50% of waking hours; 4 = Completely disabled, confined to bed or chair; 5 = Dead.
  participants
    Grade 0 | 71 | 65 | 136
    Grade 1 | 100 | 107 | 207
    Grade 2 | 18 | 16 | 34
Location of Primary Tumor [Number; unit: participants]
  Colon | 108 | 106 | 214
  Rectum | 81 | 81 | 162
  Missing | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival was defined as the time from the randomization date to the date of death. Participants who had not died by the analysis data cut-off date were censored at their last contact date and participants with survival data obtained after the planned analysis data cut-off date had survival censored at the cut-off date.
Time Frame: From randomization to the last on-study or long-term follow-up visit, as of the data cut-off date of 10 June 2014. The median follow-up time was 34.9 weeks (panitumumab plus BSC: 41.0 weeks; BSC alone: 25.5 weeks).
Population: Intent to Treat (ITT) Analysis Set (all randomized participants); participants in the ITT Analysis Set were required to have wild-type KRAS exon 2 (codons 12 and 13, alleles G12A, G12D, G12R, G12C, G12S, G12V, or G13D) per protocol.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panitumumab + BSC | BSC Alone
Number analyzed (Participants) | 189 | 188
months | 10.0 [8.7 to 11.4] | 7.4 [5.8 to 9.3]
Statistical Analysis 1: Comparison: Panitumumab + BSC vs BSC Alone; The primary hypothesis was that panitumumab plus BSC would improve overall survival compared to BSC alone. A comparison between treatments was performed using the log-rank test stratified by the randomization factors at a 5% significance level; Test type: Superiority or Other; p = 0.0096, Log Rank; Log-rank test stratified by randomization factors: geographic region (Europe vs Asia vs rest of world) and ECOG performance status (0 or 1 vs 2); Normal score = -2.59 — A normal score < 0 indicates fewer than expected events for the panitumumab plus BSC arm and therefore a longer time to event

2. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) was defined as the time from the randomization date to the date of disease progression per Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1 or death. Progressive disease (PD): At least a 20% increase in the size of target lesions compared with the smallest size since treatment started and an absolute increase of at least 5 mm, any new lesions or an increase in size of non-target lesions thought be ≥ 20% and an absolute increase of at least 5 mm, or significant increase in pleural effusions, ascites or other fluid collections with cytologic proof of malignancy. Participants who were alive and did not meet the criteria for progression by the analysis data cut-off date were censored at their last evaluable disease assessment date.
Time Frame: as for outcome 1
Population: ITT Analysis Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panitumumab + BSC | BSC Alone
Number analyzed (Participants) | 189 | 188
months | 3.6 [3.4 to 5.3] | 1.7 [1.6 to 1.9]
Statistical Analysis 1: Comparison: Panitumumab + BSC vs BSC Alone; PFS in the ITT Analysis Set was tested at a significance level of 5% conditional on a significant treatment effect on overall survival in the ITT Analysis Set; Test type: Superiority or Other; p < 0.0001, Log Rank; [statistical method as in outcome 1, analysis 1]; Normal score = -6.08 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Overall Survival in Participants With Wild-type RAS
Description: A secondary efficacy endpoint was overall survival in participants with wild-type rat sarcoma viral oncogene homolog (RAS) (without mutation in exons 2 [codons 12 and 13], 3 [codons 59 and 61], and 4 [codons 117 and 146] of KRAS and neuroblastoma RAS viral oncogene (NRAS)). In participants with wild-type RAS, RAS mutation status was defined by KRAS exon 2 mutation status per clinical trial assay testing and mutation status of KRAS exon 3 and 4 and NRAS exons 2, 3 and 4 per Sanger bi-directional sequencing. Overall survival was defined as the time from the randomization date to the date of death. Participants who had not died by the analysis data cut-off date were censored at their last contact date and participants with survival data obtained after the planned analysis data cut-off date had survival censored at the cut-off date.
Time Frame: From randomization to the last on-study or long-term follow-up visit, as of the data cut-off date of 10 June 2014. The median follow-up time was 36.1 weeks (panitumumab plus BSC: 43.7 weeks; BSC alone: 23.6 weeks).
Population: Wild-type RAS Efficacy Analysis Set (subset of participants in the ITT Analysis Set without mutation in exon 2, 3, and 4 of KRAS or NRAS)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panitumumab + BSC | BSC Alone
Number analyzed (Participants) | 142 | 128
months | 10.0 [8.7 to 11.6] | 6.9 [5.2 to 7.9]
Statistical Analysis 1: Comparison: Panitumumab + BSC vs BSC Alone; Overall survival in the Wild-type RAS Efficacy Analysis Set was compared at a significance level of 5% conditional on a significant treatment effect for progression-free survival in the ITT Analysis Set; Test type: Superiority or Other; p = 0.0135, Log Rank; [statistical method as in outcome 1, analysis 1]; Normal score = -2.47 — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Progression Free Survival (PFS) in Participants With Wild-type RAS
Description: PFS was defined as the time from the randomization date to the date of disease progression per RECIST version 1.1 or death.
  Progressive disease (PD): At least a 20% increase in the size of target lesions compared with the smallest size since treatment started and an absolute increase of at least 5 mm, any new lesions, or an increase in size of non-target lesions thought be ≥ 20% with an absolute increase of at least 5 mm, or significant increase in pleural effusions, ascites or other fluid collections with cytologic proof of malignancy. Participants who were alive and did not meet the criteria for progression by the analysis data cut-off date were censored at their last evaluable disease assessment date.
Time Frame: as for outcome 3
Population: Wild-type RAS Efficacy Analysis Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panitumumab + BSC | BSC Alone
Number analyzed (Participants) | 142 | 128
months | 5.2 [3.5 to 5.3] | 1.7 [1.6 to 2.2]
Statistical Analysis 1: Comparison: Panitumumab + BSC vs BSC Alone; PFS in the Wild-type RAS Efficacy Analysis Set was to be compared at a significance level of 5% if overall survival in the wild-type RAS Efficacy Anaysis Set demonstrated a significant treatment effect; Test type: Superiority or Other; p < 0.0001, Log Rank; [statistical method as in outcome 1, analysis 1]; Normal score = -5.98 — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Objective Response Rate
Description: Objective response rate (ORR) is defined as the percentage of participants with either a complete response (CR) or partial response (PR) per RECIST version 1.1. Radiographic tumor assessments and investigator's assessment of response were performed at Week 4, Week 8, and then every 8 weeks until disease progression (radiographic or clinical progression). CR: Disappearance of all target and non-target lesions and no new lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR: At least a 30% decrease in the size of target lesions with no progression of non-target lesions and no new lesions, or, the disappearance of all target lesions with persistence of one or more non-target lesions not qualifying for either CR or PD and no new lesions.
Time Frame: Response was assessed at Week 4, Week 8, and then every 8 weeks until the data cut-off date of 10 June 2014. The median follow-up time was 34.9 weeks (panitumumab plus BSC: 41.0 weeks; BSC alone: 25.5 weeks).
Population: ITT analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Panitumumab + BSC | BSC Alone
Number analyzed (Participants) | 189 | 188
percentage of participants | 26.98 [20.80 to 33.91] | 1.60 [0.33 to 4.59]
Statistical Analysis 1: Comparison: Panitumumab + BSC vs BSC Alone; ORR was not formally tested and the p-values are descriptive only. An exact test was used to test the hypothesis that the common odds ratio for panitumumab plus BSC relative to BSC alone for the objective response is equal to 1.0 stratified by the randomization factors; Test type: Superiority or Other; p < 0.0001, Stratified exact test; Stratified by randomization factors: geographic region (Europe vs Asia vs rest of world) and ECOG performance status (0 or 1 vs 2); Odds Ratio (OR) = 24.89, 95% CI 2-sided [7.47 to 123.77] — The odds ratio is defined as the odds of having an objective response in the panitumumab plus BSC arm relative to the odds in BSC alone arm

6. Secondary Outcome: Objective Response Rate in Participants With Wild-type RAS
Description: Objective response rate is defined as the percentage of participants with either a complete response (CR) or partial response (PR) per RECIST version 1.1. Radiographic tumor assessments and investigator's assessment of response were performed at Week 4, Week 8, and then every 8 weeks until disease progression (radiographic or clinical progression). CR: Disappearance of all target and non-target lesions and no new lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR: At least a 30% decrease in the size of target lesions with no progression of non-target lesions and no new lesions, or, the disappearance of all target lesions with persistence of one or more non-target lesions not qualifying for either CR or PD and no new lesions.
Time Frame: Response was assessed at Week 4, Week 8, and then every 8 weeks until the data cut-off date of 10 June 2014. The median follow-up time was 36.1 weeks (panitumumab plus BSC: 43.7 weeks; BSC alone: 23.6 weeks).
Population: Wild-type RAS Efficacy Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Panitumumab + BSC | BSC Alone
Number analyzed (Participants) | 142 | 128
percentage of participants | 30.99 [23.50 to 39.28] | 2.34 [0.49 to 6.70]
Statistical Analysis 1: Comparison: Panitumumab + BSC vs BSC Alone; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.0001, Stratified exact test; [statistical method as in outcome 5, analysis 1]; Odds Ratio (OR) = 20.00, 95% CI 2-sided [5.89 to 101.62] — [estimate comment as in outcome 5, analysis 1]

7. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: The severity of each AE was graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 (Grade 1 = Mild; 2 = Moderate (discomfort enough to cause interference with usual activity); 3 = Severe (incapacitating with inability to work or do usual activity); 4 = Life-threatening and 5 = Fatal), with the exception of the skin-or nail-related AEs which were graded using a CTCAE version 3.0 with modifications. A serious AE was defined as an AE that met at least 1 of the following criteria: • fatal, • life-threatening, • required in-patient hospitalization or prolongation of existing hospitalization, • resulted in persistent or significant disability/incapacity, • congenital anomaly/birth defect, and/or • other medically important serious event. Treatment-related AEs (TRAEs) are those the investigator considered there was reasonable possibility that the event might have been caused by study drug.
Time Frame: From first dose until 30 days after last dose; median safety reporting periods were 4.2 months and 2.2 months for panitumumab plus BSC arm and BSC alone arm, respectively.
Population: Safety Analysis Set (all randomized participants)
Measure: Number; unit: participants
Arm/Group | Panitumumab + BSC | BSC Alone
Number analyzed (Participants) | 189 | 188
participants
  Any adverse event (AE) | 184 | 115
  AE with worst grade of 3 | 70 | 29
  AE with worst grade of 4 | 17 | 5
  AE with worst grade of 5 | 8 | 15
  Serious adverse event (SAE) | 48 | 37
  AE leading to discontinuation of panitumumab | 20 | NA — Not applicable for BSC Alone arm
  Treatment-related adverse event (TRAE) | 166 | 7
  Treatment-related AE with worst grade of 3 | 41 | 1
  Treatment-related AE with worst grade of 4 | 4 | 1
  Treatment-related AE with worst grade of 5 | 0 | 1
  Serious treatment-related AE | 2 | 3
  TRAE leading to discontinuation of panitumumab | 1 | NA — Not applicable for BSC Alone arm

8. Secondary Outcome: Maximum Post-baseline Change From Baseline in Corrected QT (QTc) Interval
Description: QT interval is a measure of the time between the start of the Q wave and the end of the T wave in the heart's electrical cycle as measured by electrocardiogram (ECG). QTc is the QT interval corrected for heart rate. To evaluate the effect of panitumumab treatment on the QTc interval length among participants treated with panitumumab, ECGs were collected at the following time points from participants randomized to panitumumab arm at a limited number of sites: Week 1 prior to the first panitumumab infusion (Baseline) and within 30 minutes following the end of the first infusion of panitumumab (Cmax), Week 7 after 3 doses of panitumumab (steady state), and at the safety follow-up visit. The ECGs were submitted for independent central review to calculate the reported QTc interval. QTc was calculated using both the Bazett correction (QTcB) and the Fridericia correction (QTcF).
Time Frame: Baseline (pre-dose), Week 1 and Week 7 (post-dose) and 4 weeks after the last dose (Safety Follow-up visit)
Population: QTc Analysis Set is defined as the subset of participants in the Safety Analysis Set who received at least one panitumumab dose and were enrolled at the limited number of sites participating in QTc evaluation and had baseline and at least 1 post-baseline QTc assessment.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Panitumumab + BSC | BSC Alone
Number analyzed (Participants) | 53 | 0
msec
  QTcF | 14.58 (13.60) |
  QTcB | 12.57 (12.15) |

ADVERSE EVENTS:
Time Frame: From first dose until 30 days after last dose; median safety reporting periods were 4.2 months and 2.2 months for panitumumab plus BSC arm and BSC alone arm, respectively.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Panitumumab Plus BSC | BSC Alone
Serious Adverse Events (participants affected / at risk) | 48/189 | 37/188
Other Adverse Events (participants affected / at risk) | 174/189 | 74/188
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab Plus BSC (N=189) | BSC Alone (N=188)
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Bone marrow toxicity (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Pyloric stenosis (Congenital, familial and genetic disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Diplopia (Eye disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 3
Anal fistula (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 3 | 1
Intestinal obstruction (Gastrointestinal disorders) | 3 | 3
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 2
General physical health deterioration (General disorders) | 0 | 3
Malaise (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 2
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Abscess (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 2 | 0
Bronchitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Lung abscess (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Colorectal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Metastases to ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain oedema (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Speech disorder (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 1 | 1
Wallenberg syndrome (Nervous system disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 1
Obstructive uropathy (Renal and urinary disorders) | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 0 | 1
Urinary tract inflammation (Renal and urinary disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab Plus BSC (N=189) | BSC Alone (N=188)
Anaemia (Blood and lymphatic system disorders) | 15 | 16
Abdominal pain (Gastrointestinal disorders) | 28 | 18
Constipation (Gastrointestinal disorders) | 15 | 12
Diarrhoea (Gastrointestinal disorders) | 25 | 7
Dyspepsia (Gastrointestinal disorders) | 10 | 2
Nausea (Gastrointestinal disorders) | 11 | 10
Stomatitis (Gastrointestinal disorders) | 12 | 0
Vomiting (Gastrointestinal disorders) | 12 | 7
Fatigue (General disorders) | 28 | 14
Pyrexia (General disorders) | 16 | 9
Conjunctivitis (Infections and infestations) | 12 | 0
Paronychia (Infections and infestations) | 27 | 0
Weight decreased (Investigations) | 13 | 4
Decreased appetite (Metabolism and nutrition disorders) | 18 | 16
Hypocalcaemia (Metabolism and nutrition disorders) | 13 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 10 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 53 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 10
Acne (Skin and subcutaneous tissue disorders) | 26 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 54 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 29 | 1
Erythema (Skin and subcutaneous tissue disorders) | 23 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 19 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 47 | 0
Rash (Skin and subcutaneous tissue disorders) | 73 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.